CLINICAL TRIAL: NCT04606251
Title: Home-Based Telerehabilitation for People With Alzheimer Disease: A Randomized Controlled Study
Brief Title: Home-Based Telerehabilitation for People With Alzheimer Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Kübra Nur Menengiç, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kübra Nur Menengiç, IUC
Record Dates: First submitted 2020-10-24; First posted 2020-10-28 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Alzheimer Disease
Keywords: Exercise Training; Cognition; Telemedicine; Telehealth
MeSH Terms: conditions — Alzheimer Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Controlled Research Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Exercise Group (Experimental): This group will consist of the subjects taken for 6 weeks of exercise.
  Interventions: Other: Exercise
- Arm 2: Control Group (No Intervention): This group will consist of the subjects who did not receive any intervention for 6 weeks and were evaluated before and after 6 weeks.

INTERVENTIONS:
Other: Exercise — The intervention to be carried out in the study consists of physical exercises for the neck, upper and lower extremities, and trunk; It is a program that includes the addition of cognitive tasks such as memory, word finding, processing during each repetition.
  Arms: Arm 1: Exercise Group

SUMMARY:
The aim of this study is to investigate the effect of a physical exercise program with cognitive tasks to be applied with telerehabilitation in Alzheimer's disease, on cognitive and physical function, ability to perform daily living activities, depression and anxiety. Secondary aim is to examine the effect of the exercise application on the care burden and well-being of caregivers.

DETAILED DESCRIPTION:
Exercise application in the study will take 6 weeks. Evaluations will be made twice, at the beginning and end of the exercise application.

Functional mobility was measured with the 5-Times Sit-and-Stand Test (5XSTS) and Timed Up and Go Test (TUG); static balance with One-Leg Stand Test; functional independence level with Functional Independence Scale (FIM); daily living activities will be evaluated with the Katz Activities of Daily Living Scale.

The general cognitive level of the cases was determined by Mini-Mental State Examination; Depressive symptoms will be measured with the Geriatric Depression Scale-Short Form, and anxiety levels will be measured with the Beck Anxiety Scale.

The care burden of caregivers will be assessed with the Zarit Care Burden Scale, and caregiver's well-being will be assessed with the Warwick-Edinburgh Mental Well-being Scale.

Primary outcome measures are Mini Mental Test, Timed Up&Go Test, and the 5-Times Sit-and-Stand Test .

ELIGIBILITY:
Inclusion Criteria:

1. Over 65 years old,
2. Diagnosed with Alzheimer's disease according to the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease (NINCDS-ADRDA) criteria,
3. Scoring between 0-2 points according to the Clinical Dementia Rating Scale (with mild-moderate dementia-related symptoms),
4. Have used any dementia medication such as cholinesterase inhibitors and memantine for at least the last month,
5. Mini Mental Test score between 13-24 points,
6. The caregiver living with is sufficient in the use of technology,
7. Cases who could understand the instructions given in Turkish were included in the study.

Exclusion Criteria:

1. Dementia with Lewy bodies, frontotemporal dementia and one of the other types of dementia,
2. Having a pulmonary, neurological, musculoskeletal or rheumatological disease that may prevent exercise,
3. Unstable medical condition (uncontrolled diabetes or hypertension, deep vein thrombosis, etc.),
4. Modified Charlson Comorbidity Index score greater than 6,
5. Receiving any rehabilitation service from an institution or person,
6. Having regular exercise habits,
7. Subjects with visual or auditory deficits or behavioral problems that would make communication difficult were not included in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Cognitive Function-Mini Mental Test | 6 weeks
  Mini Mental Test evaluates the cognitive skills. For each question of the test, the correct answer is scored as 1 point, the incorrect answer 0 point. Test is divided into two sections, the first of which requires vocal responses only and covers orientation, memory, and attention; the maximum score is 21. The second part tests ability to name, follow verbal and written commands, write a sentence spontaneously, and copy a complex polygon; the maximum score is 9.
Timed Up and Go Test | 6 weeks
  Timed Up and Go Test measure the level of functional mobility skills and, assess fall risk and balance. The time elapsed between standing up from the sitting position, walking the distance of 3 meters, coming back and sitting back on the chair is recorded. The shorter time reflect the better performance.
Physical Mobility-5 Time Sit to Stand Test | 6 weeks
  5 Time Sit to Stand Test measure the level of functional mobility skills and, assess fall risk and lower extremity strength. The test measures the time taken to stand five times from a sitting position as quickly as possible. The shorter time reflect the better performance.

SECONDARY OUTCOMES:
Balance-One Leg Stance Test | 6 weeks
  One Leg Stance Test evaluates the static balance. The time of standing unsupported on one leg with eyes open, hands beside the body is recorded. The test is finished when the patient's foot touches the ground. Longer duration indicates good balance.
Activities of Daily Living-Katz Activities of Daily Living Scale | 6 weeks
  Katz Activities of Daily Living Scale is a questionnaire that measures the ability of people to perform daily activities functionally. The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.
Depression-Geriatric Depression Scale | 6 weeks
  The Geriatric Depression Scale is a 30-item self-report measure designed to assess and screen depressive symptoms among older adults. Each item on the GDS is scored with one point for a depressive response. Items are summed to determine the total score with a maximum of 30 points. General interpretive guidelines are as follows: scores ranging from 0 to 9 indicate normal mood, scores of 10 to 19 indicate mild depressive symptoms, and scores of 20 to 30 indicate severe depressive symptoms.
Anxiety-Beck Anxiety Inventory | 6 weeks
  The beck anxiety scale is a questionnaire used to measure the anxiety levels of individuals. Respondents are asked to report the extent to which they have been bothered by each of the 21 symptoms in the week preceding their completion of the Beck Anxiety Inventory. Each symptom item has four possible answer choices: Not at All (0 point); Mildly (1 point), Moderately (2 point), and; Severely (3 point). A total score of 0-7 is interpreted as a "Minimal" level of anxiety; 8-15 as "Mild"; 16-25 as "Moderate", and; 26-63 as "Severe".
Burden-Zarit Burden Scale | 6 weeks
  The Zarit Burden Scale is a questionnaire that measures the care burden of caregivers. It contains 22 items. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always). Higher scores indicate greater burden.
Well-being-Warwick Edinburgh Mental Well-being Scale | 6 weeks
  Warwick-Edinburgh Mental Well-being Scale measures parameters such as coping with stress, being productive and beneficial. The scale is scored by summing responses to each item answered on a 1 to 5 Likert scale. The total score is obtained by summing the score for each of the 14 items. The minimum scale score is 14 and the maximum is 70. Higher scores are associated with higher levels of mental well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Menengic KN, Yeldan I, Cinar N, Sahiner TA. Effectiveness of home-based telerehabilitation in mild to moderate Alzheimer's disease: A randomised controlled study. Alzheimers Dement. 2021 Dec;17 Suppl 8:e053406. doi: 10.1002/alz.053406. PMID 34971285